CLINICAL TRIAL: NCT06729346
Title: Can Narrow-band Imaging Detect CIS/Tumor in Normally Looking Bladder Mucosa on White Light Cystoscopy During Transurethral Resection of Bladder Tumor?
Brief Title: Is the Normal Looking Bladder Mucosa on WL Cystoscopy During TURBT Really Normal and Can NBI Detect Hidden Tumor
Status: Recruiting | Type: Observational
Sponsor: Armed Forces Institute of Urology, Rawalpindi (Other)
Responsible Party: Principal Investigator, Azmat ullah, Consultant urologist, Armed Forces Institute of Urology, Rawalpindi
Other Study IDs: Trg-1/IRB/2024/023
Record Dates: First submitted 2024-12-07; First posted 2024-12-11 (Actual); Last update posted 2025-01-29 (Actual); Status verified 2024-12

CONDITIONS: Transition Cell Cancer

STUDY DESIGN:
Observational Model: Other | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

SUMMARY:
As every urologist does transurethral resection of bladder tumor. So there are instances in which the operating surgeon is not sure whether the normal-looking mucosa or the inflammatory changes are really benign or if we are missing the CIS/bladder cancer.

DETAILED DESCRIPTION:
This is basically the observational study. in which we want to clarify that the normal-looking mucosa on white light cystoscopy is normal in reality or we are missing CIS/bladder tumor.

ELIGIBILITY:
Inclusion Criteria:

any patient with bladder tumor

-

Exclusion Criteria:

* any patient whose age is less than 18 years any patient whose age is more than 75 years

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: any patient who presented with armed forces institute of urology with bladder tumor .
Sampling Method: Probability Sample
Enrollment: 100 (Estimated)
Dates: Start 2024-12-28 (Actual); Primary Completion 2025-03-30 (Estimated); Study Completion 2025-03-30 (Estimated)

PRIMARY OUTCOMES:
to prove suspicious-looking mucosa on NBI has a bladder tumor on histopathology.. | At the time of TURBT

CONTACTS AND LOCATIONS:
Overall Officials: azmat ullah, consultant urologist, Principal Investigator — armed forces institute of urology
Locations (1):
- Armed Forces Institute of Urology, Rawalpindi, Punjab Province, Pakistan

IPD SHARING:
Plan to Share IPD: Yes
Histopathology report
Supporting Information: Study Protocol, SAP
Time Frame: 01 January 2024 till 30 march 2024
Access Criteria: each and everyone